CLINICAL TRIAL: NCT05754866
Title: Transbronchial Lung Biopsy Versus Transbronchial Lung Cryobiopsy in Critically Ill Patients With Undiagnosed Acute Hypoxemic Respiratory Failure: a Multicenter Prospective Study
Brief Title: Transbronchial Lung Cryobiopsy in Undiagnosed Acute Respiratory Failure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Shiyao Wang, Attending Physician, China-Japan Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CJFH-2022-KY-194
Record Dates: First submitted 2023-02-23; First posted 2023-03-06 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Acute Respiratory Failure; Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transbronchial lung cryobiopsy (Experimental)
  Interventions: Procedure: Transbronchial lung cryobiopsy
- Transbronchial lung biopsy (Active Comparator)
  Interventions: Procedure: Transbronchial lung biopsy

INTERVENTIONS:
Procedure: Transbronchial lung cryobiopsy — Lung tissue was obtained by transbronchial lung cryobiopsy for subsequent pathology and clinical diagnosis.
  Arms: Transbronchial lung cryobiopsy
Procedure: Transbronchial lung biopsy — Lung tissue was obtained by transbronchial lung biopsy for subsequent pathology and clinical diagnosis.
  Arms: Transbronchial lung biopsy

SUMMARY:
In patients with acute hypoxemic respiratory failure whose diagnosis is not established after initial evaluation, obtaining a histopathological diagnosis may improve the patients' prognosis. In our previous retrospective-controlled study, transbronchial lung cryobiopsy (TBLC) can lead to an increased chance of establishing a diagnosis compared with transbronchial lung biopsy (TBLB), with an acceptable safety profile. Therefore, further prospective randomized controlled studies exploring whether TBLC leads to improved prognosis for such patients are warranted.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of acute hypoxemic respiratory failure
2. Routine assessments [including bronchoscopy, bronchoalveolar lavage fluid cytology and pathogenic (including pathogenic mNGS) tests, blood tests, etc.] do not clarify the etiology, or there is an unexplained disease process
3. Imaging shows a multi-lobar segmental distribution of ground glass opacity with or without consolidations
4. Patients' families agreed to participate in the study and signed an informed consent form

Exclusion Criteria:

1. Significant hemodynamic instability
2. Uncorrectable coagulopathy
3. Severe pulmonary hypertension
4. Acute coronary syndrome
5. Intermediate-high-risk acute pulmonary embolism
6. Acute phase of stroke
7. Severe emphysema
8. Aortic dissection and massive gastrointestinal bleeding
9. Other conditions that are not suitable for participation in the clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Diagnostic yield | 7 days after procedure
  The diagnostic yield of each procedure.

SECONDARY OUTCOMES:
Mortality | 28 and 60 days
  The 28-day and 60-day of patients in each group.
Incidence of procedure related adverse events | 3 days after procedure
  Procedure related death, procedure related hemodynamic and respiratory instability, airway bleeding, pneumothorax and other procedure related adverse events.
Hospital stay | up to 60 days
  Length of hospital stay including ICU and general ward of respiratory medicine.
Organ support | up to 60 days
  Length of organ support (days).

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - China-Japan Friendship Hospital, Beijing
  - The Second Xiangya Hospital, Changsha
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - The First Affiliated Hospital of Soochow University, Suzhou
  - The Sixth Hospital of Wuhan, Wuhan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou

REFERENCES:
- [Background] Gerard L, Bidoul T, Castanares-Zapatero D, Wittebole X, Lacroix V, Froidure A, Hoton D, Laterre PF. Open Lung Biopsy in Nonresolving Acute Respiratory Distress Syndrome Commonly Identifies Corticosteroid-Sensitive Pathologies, Associated With Better Outcome. Crit Care Med. 2018 Jun;46(6):907-914. doi: 10.1097/CCM.0000000000003081. PMID 29521713
- [Background] Lim SY, Suh GY, Choi JC, Koh WJ, Lim SY, Han J, Lee KS, Shim YM, Chung MP, Kim H, Kwon OJ. Usefulness of open lung biopsy in mechanically ventilated patients with undiagnosed diffuse pulmonary infiltrates: influence of comorbidities and organ dysfunction. Crit Care. 2007;11(4):R93. doi: 10.1186/cc6106. PMID 17725820
- [Background] Philipponnet C, Cassagnes L, Pereira B, Kemeny JL, Devouassoux-Shisheboran M, Lautrette A, Guerin C, Souweine B. Diagnostic yield and therapeutic impact of open lung biopsy in the critically ill patient. PLoS One. 2018 May 25;13(5):e0196795. doi: 10.1371/journal.pone.0196795. eCollection 2018. PMID 29799835
- [Background] Papazian L, Doddoli C, Chetaille B, Gernez Y, Thirion X, Roch A, Donati Y, Bonnety M, Zandotti C, Thomas P. A contributive result of open-lung biopsy improves survival in acute respiratory distress syndrome patients. Crit Care Med. 2007 Mar;35(3):755-62. doi: 10.1097/01.CCM.0000257325.88144.30. PMID 17255856
- [Background] Zhou G, Feng Y, Wang S, Zhang Y, Tian Y, Wu X, Zhao L, Wang D, Li Y, Tian Z, Zhan Q. Transbronchial lung cryobiopsy may be of value for nonresolving acute respiratory distress syndrome: case series and systematic literature review. BMC Pulm Med. 2020 Jun 29;20(1):183. doi: 10.1186/s12890-020-01203-w. PMID 32600302
- [Background] Wang S, Feng Y, Zhang Y, Tian Y, Gu S, Wu X, Feng Y, Zhao L, Liu M, Wang D, Li Y, Tian Z, Wang S, Huang X, Zhou G, Zhan Q. Transbronchial lung biopsy versus transbronchial lung cryobiopsy in critically ill patients with undiagnosed acute hypoxemic respiratory failure: a comparative study. BMC Pulm Med. 2022 May 4;22(1):177. doi: 10.1186/s12890-022-01966-4. PMID 35509092
- [Background] Wang S, Zhou G, Feng Y, Zhang Y, Tian Y, Gu S, Wu X, Li M, Feng Y, Wang D, Li Y, Tian Z, Zhao L, Li M, Chen W, Huang X, Zhan Q. Feasibility of transbronchial lung cryobiopsy in patients with veno-venous extracorporeal membrane oxygenation support. ERJ Open Res. 2022 Dec 19;8(4):00383-2022. doi: 10.1183/23120541.00383-2022. eCollection 2022 Oct. PMID 36545213
- [Background] Chang CH, Ju JS, Li SH, Wang SC, Wang CW, Lee CS, Chung FT, Hu HC, Lin SM, Huang CC. Feasibility and Safety of Transbronchial Lung Cryobiopsy for Diagnosis of Acute Respiratory Failure with Mechanical Ventilation in Intensive Care Unit. Diagnostics (Basel). 2022 Nov 23;12(12):2917. doi: 10.3390/diagnostics12122917. PMID 36552923